CLINICAL TRIAL: NCT03845959
Title: NGHIÊN CỨU NGẪU NHIÊN, MÙ ĐÔI, CÓ ĐỐI CHỨNG TRONG ĐIỀU TRỊ HỘI CHỨNG CỔ VAI CÁNH TAY CỦA VIÊN NANG CỨNG TD 0019 (A Randomized, Double Blind, Placebo Controlled, Parallel Group, Phase 3 Trial to Evaluate the Satety and Efficacy of Therapy With Hard Capsule TD0019 in Cervical Scapulohumeral Syndrome)
Brief Title: A Trial of TD0019 in Treatment of Cervical Scapulohumeral Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sao Thai Duong Joint Stock Company (Industry)
Collaborators: Big Leap Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TD0019.02
Record Dates: First submitted 2019-01-10; First posted 2019-02-19 (Actual); Last update posted 2019-02-19 (Actual); Status verified 2018-02

CONDITIONS: Syndrome Pain
MeSH Terms: conditions — Somatoform Disorders

STUDY DESIGN:
Intervention Model Description: Three arms: basic dose, 1.5 basic dose and placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TD0019.6cap (Experimental): estimated dose, 2 oral capsules/time x 3 times/day
  Interventions: Drug: TD0019 oral capsule
- TD0019.9cap (Experimental): 1.5 times of estimated dose 2 oral capsules/time x 3 times/day
  Interventions: Drug: TD0019 oral capsule
- Placebo (Placebo Comparator): Placebo 2 placebo oral capsules /time x 3 times/day
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: TD0019 oral capsule — TD0019 are green, hard capsule with size 0, containing yellow herbal powder with special smell of herbal.
  Other Names: Vien Vai Gay Thai Duong
  Arms: TD0019.6cap; TD0019.9cap
Drug: Placebo oral capsule — Placebo
  Arms: Placebo

SUMMARY:
Cervical scapulohumeral syndrome, which is also called scapulohumeral syndrome or cervical radiculopathy is a group of syndromes related to cervical spine disorders with disfunctional nerves and without inflamation. The physical syndromes vary from neck pain, Sensory Processing Disorder/Movenment Disorder of areas dominated by injured nerves.

The hard capsule TD0019 is a product based on the traditional prescription named "Độc hoạt tang ký sinh thang" combined with Nattokinase and the extraction of Salix alba Cortex

.

DETAILED DESCRIPTION:
Cervical scapulohumeral syndrome, which is also called scapulohumeral syndrome or cervical radiculopathy is a group of syndromes related to cervical spine disorders with disfunctional nerves and without inflamation. The physical syndromes vary from neck pain, hands, accompanied by a Sensory Processing Disorder/Movenment Disorder of areas dominated by injured nerves. The most common reason is Cervical spondylosis The hard capsule TD0019 is a product based on the traditional prescription named "Độc hoạt tang ký sinh thang" combined with Nattokinase and the extraction of Salix alba Cortex.

The trial lasts for 24 months with 4 subject visits (from T0 to T3) and is conducted in National Hospital of Traditional Medicine (Hanoi, Vietnam).

Screening procedure occurs at T0 visit, followed by T1 (15+-3 days) and T2 (30+-3 days).

There are 2 levels of dosages: basic dose (arm 1) and 1.5x (arm 2) of basic dose.

There is also another arm using placebo, thus the trial have 3 arms in total.

ELIGIBILITY:
Inclusion Criteria:

Subject must meet all below criteria to be enrolled:

* Subjects diagnosed with cervical scapulohumeral syndrome according to the Guideline of Vietnam MOH 2014
* Age > 18 at time of signing ICF, male or female.
* No contraindications with oral NSAIDs.
* Agree and and sign in the ICF

Exclusion Criteria:

Subjects will be excluded in the trial if any of the below are met:

* Hypersensitivity to any subtances of TD0019 or any NSAIDs.
* Pregnant or lactating.
* Currently having surgical indications.
* Movement disorders, diabetes, myasthenia, alcoholism
* Other conditions asseted by the investigator that are not eligible to be enrolled.
* Cervical scapulohumeral syndrome caused by tumor, infection, hypertension, physical injured.
* Arrhythmia, hypertension.
* Hypertensitivity to meloxicam or its excipients.
* Cross - hypertensitivity to aspirin or other NSAIDs.
* Peptic ulcer
* Severe liver failure
* Severe renal failure without dialysis.
* Gastrointestinal hemorrhage, recent brain hemorrhage.
* Uncontrolled heart failure.
* Alcoholism, movement disorders, diabetes, muscular dystrophy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2017-08-30 (Actual); Primary Completion 2017-12-20 (Actual); Study Completion 2018-02-20 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Pain Scores on the Visual Analog Scale at day 15th, day 30th, 1 month after end of study. | day 15th, day 30th, 1 month after end of study.
  VAS scale: 0 = no pain | 0-->2: mild | 2-->4: moderate | 4--> 6: severe | 6->8: extreme | 8-->10: untolerable
Change in Range of Motion of cervical spine | day 15th, day 30th, 1 month after end of study.
  Analog and traditional devices to measure range of motion in the joints of the body include the goniometer and inclinometer which use a stationary arm, protractor, fulcrum, and movement arm to measure angle from axis of the joint.
Change in symptoms of nerve root compression | day 15th, day 30th, 1 month after end of study.
  The presence of numbness or weakness of the buttock and leg
Change in limitation of daily rountines | day 15th, day 30th, 1 month after end of study.
  Neck Disability Index at day 15th, day 30th, 1 month after end of study.
Frequency of AE, SAE. | 1 month
  CTCAE 4.0

CONTACTS AND LOCATIONS:
Locations (1):
- National Hospital of Traditional Medicine, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No